CLINICAL TRIAL: NCT04351919
Title: Assessment of Efficacy and Safety of HCQ and Antibiotics Administrated to Patients COVID19(+), inTunisia
Brief Title: Assessment of Efficacy and Safety of HCQ and Antibiotics Administrated to Patients COVID19(+)
Acronym: COVID+PA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: - Interest in the use of HCQ is controversial.
Sponsor: Abderrahmane Mami Hospital (Other)
Collaborators: Eshmoun Clinical Research Center (Network); Dacima Consulting (Other)
Responsible Party: Principal Investigator, Dr Jalila Ben Khelil, Head of department, Abderrahmane Mami Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECC2020-04
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Patients With COVID19
MeSH Terms: interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Intervention Model Description: open, interventional, multicentric study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCQ Arm (Experimental)
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine — 400mg per day during 10 days
Drug: Azithromycin — 500 mg per day during 5 days

SUMMARY:
The study will assess the number of patients who become asymptomatic from clinical signs of COVID19 and will assess the efficacy of Hydroxychloroquine (HCQ) and Azithromycine effects on paucisymptomatic patients with ou without co-morbidities

ELIGIBILITY:
Inclusion Criteria:

* confirmed COVID19 (+)
* Qt<500ms
* no severity criteria
* pauci-symptomatique patients
* signed consent form

Exclusion Criteria:

* no confirmed patient COVID19
* severity criteria
* known allegies to macrolides and HCQ
* Treated with HCQ within 1 month prior to inclusion
* hepatitis insufficiency
* Renal insufficiency
* treatment no indicated with azithro and HCQ
* hypovolemia
* complete brach block
* retinopathia
* psoriasis
* pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-05 (Estimated); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
improvment or healing of clinical signs | at the end of the study treatment - 1 month after inclusion
  no respiratory infectious signs
Evolution of clinical signs | at the end of the study treatment - 1 month after inclusion
  Low respiratory signs with severity criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Eshmoun Clinical Research Centre/ Hôpital Abderrahmen Mami-Ariana, Tunis, Tunisia